CLINICAL TRIAL: NCT03764098
Title: Mechanistic Evaluation of Guanfacine on Drinking Behavior in Women and Men With Alcohol Use Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000023970; P01AA027473 (NIH); U54AA027989 (NIH)
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use
MeSH Terms: conditions — Alcohol Drinking | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guanfacine ER (Experimental): Guanfacine extended release (6mg/day ER). Administered orally twice daily at 8:00 AM and 8:00 PM while titrating to the full dose. Titration schedule: Days 1-3 1mg/day; 0.5mg/dose, Days 4-6 2mg/day; 1mg/dose, Days 7-9 3mg/day; 1.5mg/dose, Days 10-12 4mg/day; 2mg/dose; Days 13-15 5mg/day; 2.5mg/dose and Days 16-23 6mg/day; 3mg/dose. Once at steady state, administration is orally once per day at 8:00 PM.
  Interventions: Drug: Guanfacine ER
- Placebo (Placebo Comparator): Administered orally twice a day at 8:00 AM and 8:00 PM Days 1-23, then orally once a day at 8:00 PM.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Guanfacine ER — Guanfacine Extended Release (6mg/day ER)
  Other Names: Intuniv
  Arms: Guanfacine ER
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
For this protocol, the investigators plan to collect pilot data to examine sex differences in guanfacine's effect on 1) counteracting stress and stimulation based drinking behavior in the laboratory and 2) improving clinical outcomes during a subsequent treatment phase.

DETAILED DESCRIPTION:
This study is a double blind, placebo controlled, parallel group design, which will compare guanfacine (6mg/day ER) to placebo (0mg/day) in treatment seeking adults meeting criteria for DSM V alcohol use disorders (160, 40 per med x sex cell).

Eligibility screening consists of an intake session and a physical exam. Subjects meeting eligibility criteria will be randomized to 6mg/day ER guanfacine or matching placebo, stratified by sex. Titration to steady state medication levels will occur over a 3 week period (Weeks minus 3 to minus 1). Subjects will then complete three laboratory sessions during Week 0 to evaluate ad lib consumption.

During each laboratory session, personalized imagery (within subject factor, stress, stimulating, or neutral/relaxing, order balanced) will precede a 2 hour alcohol self-administration period. Subjects will then begin a 6 week treatment phase (Week 1 to 6) where medication is combined with a medical management platform delivered at weekly appointments.

At the end of the treatment phase, medication will be tapered for 5 days, and a final follow up evaluation will occur 1 and 3 months following the end of treatment. Primary outcome measures include the number of drinks consumed during the three self-administration sessions, and reduction in percent heavy days of drinking during treatment.

Adverse events are evaluated at each study appointment and will be tabulated. The date March 1, 2019 was used as the actual start date that was associated with the preliminary funding. The study start date has been updated to reflect the beginning of the U54 grant.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 70;
2. Able to read and write English;
3. Meets DSM V criteria for current (past 6 months) alcohol use disorder or Drinking criteria: Males Drinks more than 14 drinks per week and exceeds 4 drinks per day at least twice per week; Females Drinks > more than 7 drinks per week and exceeds 3 drinks per day at least twice per week. Must meet drinking criteria during a consecutive 30 day period prior to baseline;
4. Laboratory sessions will be scheduled such that subjects will not have major responsibilities on the following day which might limit drinking during the self administration session (e.g., job interview, exam);
5. Able to take oral medications and willing to adhere to medication regimen;
6. indicate willingness to cut down on drinking during the treatment period.

Exclusion Criteria:

1. Subjects with any significant current medical conditions (neurological, cardiovascular [including hypertension or hypotension: sitting BP more than 160/100 or less than 90/60mmHg at baseline screening], endocrine, thyroid, renal, liver), seizures, delirium or hallucinations, or other unstable medical conditions including HIV;
2. Current DSM V substance use disorder, other than alcohol abuse disorder or nicotine dependence;
3. A positive test result at intake appointment on urine drug screens conducted for illicit drugs;
4. Past 30 day use of psychoactive drugs including anxiolytics and antidepressants;
5. Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD);
6. Suicidal, homicidal or evidence of current (past 6 month) mental illness such as schizophrenia, bipolar disorder or major depression, or anxiety disorders;
7. Meet DSM V criteria for current (past 6 month) ADHD;
8. Only one member per household can participate in the study
9. Specific exclusions for administration of guanfacine not already specified include: EKG evidence at baseline screening of any clinically significant conduction abnormalities or arrhythmias; known intolerance for guanfacine or any alpha blocker; history of fainting, syncopal attacks, heart failure or myocardial infarction, or impaired liver (AST, ALT > 3x normal) or renal function (estimated creatinine clearance <60 cc/min); treatment with any antihypertensive drug or any alpha adrenergic blocker; use of any CNS depressant (e.g., phenothiazines, barbiturates, benzodiazepines);
10. Subjects likely to exhibit clinically significant alcohol withdrawal during the study. Specifically, we will exclude subjects who a) have a history of perceptual distortions, seizures, delirium, or hallucinations upon withdrawal, or b) have a score of more than 8 on the Clinical Institute Withdrawal Assessment scale at intake appointments;
11. Subjects who have taken any investigational drug within 4 weeks immediately preceding admission to the treatment period;
12. Participation within the past 8 weeks in other studies that involve additive blood sampling and/or interventional measures that would be considered excessive in combination with the current application;
13. at intake express desire to completely abstain from alcohol;
14. currently in treatment for alcohol use

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption | 120 minutes
  Means mls of alcohol consumed for guanfacine ER and placebo groups during 120 minute alcohol self administration sessions with personalized stress imagery vs stimulation imagery vs neutral imagery taking place as close to Week 0 of steady state as possible comparing females to males.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No